CLINICAL TRIAL: NCT05884580
Title: Neuflo Water Electrolysis System for the Treatment of Benign Prostatic Hyperplasia
Brief Title: Neuflo System for the Treatment of BPH
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: A design change was required following the first treatment. The design concept was not feasible.
Sponsor: ProstaCare Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Neuflo-CIP-ANZ-202303
Record Dates: First submitted 2023-05-23; First posted 2023-06-01 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: prostate; catheter; IPSS
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, single-arm clinical evaluation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants receiving treatment with the Neuflo BPH Treatment System. (Experimental)
  Interventions: Device: Neuflo BPH Treatment System

INTERVENTIONS:
Device: Neuflo BPH Treatment System — The Neuflo BPH Treatment System is designed to treat patients with lower urinary tract symptoms (LUTS) associated with BPH. It is an outpatient-based, minimally invasive treatment option and uses hydrolysis to reduce prostatic tissue in the lateral lobes of the prostate. Reduced pressure and constriction of the urethra alleviates urinary and other symptoms of BPH.
  Other Names: Neuflo Water Hydrolysis System

SUMMARY:
The goal of this clinical study is to assess the effectiveness and safety of the Neuflo System for the treatment of benign prostatic hyperplasia (BPH). The main questions it aims to answer are:

* Can treatment with the Neuflo System lead to at least a 30% improvement in lower urinary tract symptoms (LUTS) secondary to BPH, as measured by the international prostate symptom score (IPSS) at 3 months after treatment which is sustained for 12 months?
* Is treatment with the Neuflo System tolerable to the patient, as measured by visual analog score (VAS) for pain before and after treatment and procedural medication requirements?
* Is treatment with the Neuflo System safe, as measured by the incidence and severity of device or procedural related serious adverse events.

Participants will be enrolled in the study over a 6 month period. Each participant will be treated with the Neuflo System and assessed at 3 and 12 months following treatment. A subgroup of patients will have an MRI at 1 week to assess the volume and location of ablated tissue.

The duration of the study is expected to be 18 months.

DETAILED DESCRIPTION:
This is a prospective, multicentre, single-arm clinical study in a sample of up to 25 participants across study sites in Australia and New Zealand. The aim of the study is to assess the effectiveness and safety of treatment with the Neuflo BPH Treatment System to relieve lower urinary tract symptoms (LUTS) secondary to benign prostatic hyperplasia (BPH).

BPH is characterised by the benign growth of stromal and epithelial cells around the prostatic urethra causing obstruction and LUTS which include urinary retention, frequent urination, dysuria, nocturia, and increased risk of urinary tract infections. Although BPH is a benign condition, the resulting symptoms can greatly reduce quality of life.

The Neuflo System uses water electrolysis and the associated changes in pH to ablate the prostate cells in the region surrounding electrodes which are placed into the tissue via the urethra. The shaft of the Neuflo device is inserted by the clinician into the urethra within a Foley catheter which has been anchored in the bladder. The device is operated using a handle attached to a battery-powered control unit which provides a low level charge. When the tip of the shaft is positioned adjacent to the prostate, the clinician deploys four small electrodes which move through the Foley catheter and urethral wall into the prostate. The clinician then starts the treatment using the Control Unit. The Control Unit delivers a defined current for a defined duration and turns off automatically. The electrodes are then retracted and the device removed. The Foley catheter may be removed or remain according to clinical needs.

The treatment process is not expected to cause any more than mild discomfort and be completed within 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all inclusion criteria to participate in this study.

1. Males aged 45 years of age or older
2. IPSS score of 13 or higher
3. Eligible uroflow with unadjusted or adjusted peak flow rate of equal to or less than 13ml/sec with a corresponding:

   1. voided volume of at least 100 ml, and,
   2. Post Void Residual (PVR) of 250 ml or less
4. Prostate volume of 25-80 cm3, inclusive as measured by ultrasound or MRI
5. Prostatic sagittal length of 3.2 cm or greater, as measured by ultrasound or MRI
6. Prostatic transverse width of 3.5 cm or greater as measured by ultrasound or MRI
7. Prostatic anterior-posterior height of 2.5 cm or greater as measured by ultrasound or MRI
8. Participant must have the ability to understand and consent to participate in this study
9. Participant must be willing and able to participate in follow-up evaluations

Exclusion Criteria:

Participants meeting any of the exclusion criteria listed at baseline will be excluded from participation.

1. Outlet obstruction due to an enlarged middle lobe or significant central gland of the prostate
2. Significant transverse asymmetry of prostatic lateral lobes
3. Participant has an implantable pacemaker or cardiac defibrillator
4. Participant has a penile implant
5. History or current diagnosis of prostate cancer or bladder cancer
6. Active urinary tract infection (UTI) (Note: participant can be enrolled if the UTI is treated and followed with a negative urine test result)
7. Neurogenic, decompensated, or atonic bladder
8. Overactive bladder in the absence of prostatic obstruction
9. Current, recurrent (two or more) urethral strictures or muscle spasms that prevent insertion of the catheter
10. Bleeding disorders or takes anticoagulation medications unless anti-platelet medication has been discontinued for at least 7 days prior to treatment (Participants are allowed to delay or repeat screening to fulfil this requirement)
11. Previous rectal surgery other than haemorrhoidectomy
12. Previous radical pelvic surgery or pelvic irradiation
13. Interest in maintaining fertility
14. Previous surgery or minimally invasive procedure(s) to treat symptomatic BPH
15. Use of Alpha blocker for the treatment of BPH within 14 days of treatment date. (Participants are allowed to delay or repeat screening to fulfil this requirement)
16. 5-ARI (5-alpha-reductase inhibitor), (an enzyme inhibitor) use within 3 months of treatment date (Participants are allowed to delay screening to fulfil this requirement)
17. Concomitant bladder stones
18. History of other diseases or conditions causing voiding dysfunction
19. Current medication affecting bladder function
20. Known allergy to nickel
21. Chronic prostatitis, recurrent prostatitis, chronic pelvic pain syndrome (CPPS), or painful bladder syndrome within the past 12 months
22. History of medical, surgical, or other conditions that, in the opinion of the investigator, would limit study participation

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-11-10 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-10 (Actual)

PRIMARY OUTCOMES:
Effectiveness: Relief of BPH symptoms as measured by International Prostate Symptom Score (IPSS) | 3 months after treatment
  Participants IPSS scores have a possible range of 13 to 35 with higher scores indicating more severe symptoms. Effective relief of BPH symptoms will be indicated by improvement (reduction) at 3 months of at least 30% from baseline IPSS score.

SECONDARY OUTCOMES:
Improvement in urinary function (Qmax) | At 3 months after treatment
  Urinary Flow rate is measured in ml per second with higher flow rate indicating superior urinary function. Improvement in urinary function will be indicated by increased Maximum Flow Rate (Qmax) at 3 months relative to baseline.
Improvement in urinary function (PVR) | At 3 months after treatment
  Post Void Residual (PVR) is a measure of the amount of urine left in the bladder after a voluntary void and is measured in ml. Improvement in urinary function will be indicated by reduced PVR at 3 months relative to baseline.
Improvement in sexual function | At 3 months after treatment
  Sexual function will be measured using the International Index of Erectile Function (IIEF) where lower scores indicate worse erectile dysfunction. Improvement in sexual function will be indicated by higher scores on the IIEF at 3 months relative to baseline.
Improvement in quality of life | At 3 months after treatment
  Quality of Life due to urinary symptoms (QoL) measured on a scale of 0 to 7 with higher scores indicating worse quality of life. Improvement in QoL indicated by a lower score at 3 months relative to baseline.
Treatment tolerability & procedural medication requirements | On day of treatment only
  Visual Analog Scale (VAS) to measure pain before, during, and immediately following treatment. VAS to measure pain from 0 to 10 with higher scores indicating more pain. Procedural medication requirements to be captured in instances where medication is used.
Secondary intervention and medication use for Lower Urinary Tract Symptoms (LUTS) | At 3, 6 and12 months after treatment
  Document use of secondary intervention for treatment of LUTS and medication requirements at follow up visits beyond 6 weeks.
Neuflo System performance | On day of treatment only
  Frequency of system deficiencies including adverse events during treatment.
Neuflo System performance on Larger Prostates | At 3 months after treatment
  Comparison of primary outcome on 56cm3 to 80cm3 prostates relative to 25cm3 to 55cm3 prostates
Maintenance of improvement of LUTS | At 12 months after treatment
  Percent change in IPSS score between baseline and 12 months after treatment.
Participant satisfaction | 1 and 6 weeks, and 3, 6 and 12 months after treatment
  Participant satisfaction score (satisfied with the procedure) measured on a 5 point scale with higher scores indicating greater satisfaction.

OTHER OUTCOMES:
Safety: safety of the Neuflo System | Up to 12 months after treatment
  Incidence and severity of device and/or procedural serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Bay of Plenty, Tauranga, Tauranga, New Zealand

IPD SHARING:
Plan to Share IPD: No